CLINICAL TRIAL: NCT04600232
Title: Clinical Utility of TB-LAM in the Diagnosis of Active TB in Hospitalized HIV-infected Patients
Brief Title: TB-LAM in the Diagnosis of TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Jun Chen, Shanghai Public Health Clinical Center, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TB-LAM
Record Dates: First submitted 2020-10-20; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections; Tuberculosis; Non-Tuberculous Mycobacterial Pneumonia
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnosis arm (Experimental): Urine TB-LAM, sputum smear, Gene Xpert, mycobacterial culture
  Interventions: Diagnostic Test: Alere TB-LAM

INTERVENTIONS:
Diagnostic Test: Alere TB-LAM — Subjects also undergo clinical evaluation including CT, sputum smear, Gene Xpert and mycobacterial culture.

SUMMARY:
Tuberculosis (TB) is still the leading cause of death in HIV-infected patients. Early diagnosis of TB substantially improves the survival of HIV-infected patients. Urine based detection of lipoarabinomannan (LAM) provides promising methods for quick diagnosis of TB in HIV-infected patients. However, the sensitivity and specificity of TB-LAM is still not well established, especially in area where non-tuberculosis mycobacterium is also prevalence. Here we aimed to evaluate the clinical utility of TB-LAM in diagnosis of active TB in hospitalized HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized HIV-infected patients.
* Willing to participate into the study.

Exclusion Criteria:

* Already diagnosed with active TB
* Received any anti-tuberculosis drugs and/or quinolone for more than 7 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity against microbiological reference standard | 2 months
  Number of TB-LAM positive/Number of positive by culture or Gene Xpert
Specificity against microbiological reference standard | 2 months
  1-Number of TB-LAM negative/Number of negative by culture or Gene Xpert or smear

SECONDARY OUTCOMES:
Sensitivity against composite reference standard | 2 months
  Number of TB-LAM positive/Number of active TB diagnosed clinically
Specificity against composite reference standard | 2 months
  1-Number of TB-LAM negative/Number of TB excluded

IPD SHARING:
Plan to Share IPD: No
Participant data without individual identification can be provided upon request.